CLINICAL TRIAL: NCT01658449
Title: Comparison of the Tolerability of Two Formulations of Hypertonic Saline in Cystic Fibrosis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ospedale Civile Ca' Foncello (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: HS/2009 HYANEB
Record Dates: First submitted 2012-07-13; First posted 2012-08-07 (Estimated); Last update posted 2012-08-10 (Estimated); Status verified 2009-02

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- group A (Experimental)
  Interventions: Other: Inhalable Hypertonic saline 7% + Hyaluronan 0.1%
- group B (Experimental)
  Interventions: Other: Inhalable Hypertonic saline 7%

INTERVENTIONS:
Other: Inhalable Hypertonic saline 7% + Hyaluronan 0.1% — Administration of Inhalable Hypertonic saline 7% + Hyaluronan 0.1% 5 ml twice a day, after bronchodilator for one month.
  Arms: group A
Other: Inhalable Hypertonic saline 7% — Administration of Inhalable Hypertonic saline 7% 5 ml twice a day, after bronchodilator for one month.
  Arms: group B

SUMMARY:
The purpose of this study is to compare the tolerability and acceptability of a formulation containing Hypertonic saline 7% (HS) alone and a formulation containing HS and Hyaluronic acid 0.1% in a population of Cystic Fibrosis (CF) patients who already showed poor tolerance to HS.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of Cystic Fibrosis (genotyping and sweat test)
* > 8 year-old
* clinically and therapeutically stable disease in the last 30 days;
* Forced Expiratory Volume in one second (FEV1) ≥ 50% of predicted value;
* intolerance (cough, throat irritation, saltiness) to previous administration of 5.8% hypertonic saline solution.

Exclusion Criteria:

* decrease in FEV1 >15% after first inhalation of hypertonic saline;
* Burkholderia cepacia infection;
* infective exacerbation requiring antibiotic treatment in the 15 days preceding enrolment;
* patient non compliant to standard therapy;
* Lung transplant;
* Patient unable to perform reproducible spirometry;
* Intolerance to β2 bronchodilators;
* Concurrent enrolment in other clinical trials;
* Plasmatic creatinine and transaminases more than twice the normal values.

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-12; Primary Completion 2011-06 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Comparison of the judgement on global pleasure of the inhalation between the two treatment groups | The outcome measure was assessed at day 1, day 7, day 14, day 21, and day 28 of the four-weeks treatment period. For each time-point we operated a comparison between the two groups.
  A judgment on acceptability and global pleasure of the inhalation was weekly reported by patients on a diary, expressed on a 1-10 scale: a score lower than 6 was considered unfavourable.
Comparison of the symptom cough between the two treatment groups | The outcome measure was assessed at day 1, day 7, day 14, day 21, and day 28 of the four-weeks treatment period. For each time-point we operated a comparison between the two groups.
  A judgement on the symptom cough, one of the most important causes of HS intolerance and poor compliance to HS treatment, was weekly reported by patients on a diary, as assessed on a scale of four grades (absent, mild, moderate, severe).
Comparison of the sensation of saltiness between the two treatment groups | The outcome measure was assessed at day 1, day 7, day 14, day 21, and day 28 of the four-weeks treatment period. For each time-point we operated a comparison between the two groups.
  A judgement on the sensation of saltiness, one of the most important causes of HS intolerance and poor compliance to HS treatment, was weekly reported by patients on a diary, as assessed on a scale of four grades (absent, mild, moderate, severe).
Comparison of the sensation of throat irritation between the two treatment groups | The outcome measure was assessed at day 1, day 7, day 14, day 21, and day 28 of the four-weeks treatment period. For each time-point we operated a comparison between the two groups.
  A judgement on the sensation of throat irritation, one of the most important causes of HS intolerance and poor compliance to HS treatment, was weekly reported by patients on a diary, as assessed on a scale of four grades (absent, mild, moderate, severe).

SECONDARY OUTCOMES:
Comparison of Delta FEV1 between the two treatment groups | day 1 and day 28 of the four-weeks treatment
  Secondary outcome was the effect on respiratory function. A sequence of spirometries was performed as follows. A spirometry was performed in basal conditions, then 400 ug of salbutamol were administered and spirometry was performed again after 15 minutes. Whitin 30 minutes, the first dose of the randomized formulation was administered for 15 minutes and a third spirometry was performed 30 minutes after the inhalation. This sequence was repeated 4 weeks later, with the administration of the last dose of treatment.
  Delta FEV1 was calculated as follows: [(FEV1 after randomized solution inhalation - FEV1 after bronchodilator)/FEV1 after bronchodilator]x 100. Delta FEV1 was the outcome measure used to compare the two groups of treatment both at the first dose of the four-weeks treatment and at the end (last dose)of the four-weeks treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- centro Fibrosi Cistica, Treviso, Italy, Italy

REFERENCES:
- [Derived] Ros M, Casciaro R, Lucca F, Troiani P, Salonini E, Favilli F, Quattrucci S, Sher D, Assael BM. Hyaluronic acid improves the tolerability of hypertonic saline in the chronic treatment of cystic fibrosis patients: a multicenter, randomized, controlled clinical trial. J Aerosol Med Pulm Drug Deliv. 2014 Apr;27(2):133-7. doi: 10.1089/jamp.2012.1034. Epub 2013 Jun 8. PMID 23745525